CLINICAL TRIAL: NCT01829451
Title: Autocrosslinked Hyaluronic Acid Gel in Prevention of Intrauterine Adhesions After Bipolar Radiofrequency Endometrial Ablation: a Randomised, Controlled and Double Blind Study
Brief Title: Hyaluronic Acid Gel in Prevention of Intrauterine Adhesions After Endometrial Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Uoulu
Record Dates: First submitted 2013-03-14; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic acid gel (Experimental): Hyaluronic acid gel is placed into the uterus after endometrial ablation
  Interventions: Other: Hyaluronic acid gel
- No hyaluronic acid gel (Placebo Comparator): An empty Pipelle device is taken into the uterus after endometrial ablation as an placebo procedure

INTERVENTIONS:
Other: Hyaluronic acid gel — Hyaluronic acid gel is placed into the uterus after endometrial ablation
  --------------------------------------------------------------------------------
  Arms: Hyaluronic acid gel

SUMMARY:
The aim of the study is to evaluate if hyaluronic acid gel prevents intrauterine adhesion formation after endometrial thermal ablation.

ELIGIBILITY:
Inclusion Criteria:

* menorrhagia

Exclusion Criteria:

* abnormal uterine cavity,
* abnormal endometrial biopsy

Ages: 35 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
prevention of intrauterine adhesion formation | 3 months
  The effect of hyaluronic acid gel on the formation of intrauterine adhesions after endometrial thermal ablation is assessed in an outpatient hysteroscopy after 3 months. Classification of intrauterine adhesions has been created for this study specifically.